CLINICAL TRIAL: NCT07321353
Title: Online Problem-Solving Intervention for Brain Tumor Survivors: A Two-site, Two-arm Pilot Randomized Controlled Trial
Brief Title: Survivors Journey+
Acronym: SJ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0546; HT9425-24-1-0746 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-07

CONDITIONS: Pediatric Brain Tumor
Keywords: pediatric brain tumor survivors; online learning; Adolescent young adult; Family; Digital; Problem Solving

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Survivors Journey Program (Experimental): The Survivor's Journey+ (SJ+) intervention seeks to address "gaps in quality of life and/or survivorship that may impact mission readiness and the health and well-being of military members, Veterans, their beneficiaries, and the general public" by providing training in stress management, problem-solving, metacognitive strategies, self-regulation, and communication in the context of a contextualized, developmentally tailored intervention to address the multifaceted challenges facing adolescent/emerging adult PBTS and their families.
  Interventions: Behavioral: Survivor's Journey+
- Internet Resources Comparison (Experimental): IRC families will receive access to a home page of pediatric brain tumor survivor resources and links (identical to those given on the SJ+ homepage) but will not be able to access specific session content. This will enable us to equate the groups with respect to access to the information and resources available on the Web.
  Interventions: Behavioral: Survivor's Journey+

INTERVENTIONS:
Behavioral: Survivor's Journey+ — Our overarching objectives are to: 1) to refine the existing program based on feedback from patient advocates and establish usability and accessibility; 2) examine the efficacy of SJ+ in improving global QoL, internalizing symptoms, and EF skills in adolescent/emerging adult PBTS; and 3) examine the efficacy of SJ+ in reducing caregiver depression and family impact.
  Other Names: SJ+

SUMMARY:
The main goal of this pilot randomized controlled trial is to learn if an online program called "Survivors Journey" (SJ+) can help teens and young adults, ages 15-25, who are Pediatric Brain Tumor Survivors (PBTS), and their caregivers, manage everyday challenges better by using skills like problem-solving and coping skills. The main questions it aims to answer are:

* Is the SJ+ program rated as feasible (>50% enrollment rate and >75% retention rate) and acceptable (>80% satisfaction rate) by PBTS and their caregivers?
* Does the SJ+ program have better outcomes in improving PBTS and caregiver wellbeing in comparison to an internet resource comparison (IRB) made for PBTS and their families? Participants will be randomized into two groups: one group will be given access to the online SJ+ program and receive weekly online coaching sessions, and the other group will be given access to an IRC. Outcomes will be assessed at baseline, treatment completion (~ 3 months post-baseline), and at follow-up six months post-baseline. These outcomes include quality of life, internalizing symptoms, performance-based executive function skills, depression, and family impact.

DETAILED DESCRIPTION:
Pediatric brain tumor survivors (PBTS) experience worse outcomes compared to other survivors or healthy adolescents and young adults. This includes quality of life (QoL), neurocognitive late effects, declines in IQ, executive functioning (EF), and social problem-solving skills. As adolescents navigate academic and social challenges, neurocognitive late effects place PBTS at elevated risk for impaired functioning during this critical transition. Equipping PBTS and their caregivers with a set of skills to manage stress, solve problems, and address neurocognitive and social challenges may promote better outcomes and prevent further declines in QoL. Prior research has targeted the survivor or caregiver in isolation, and not as family-centered treatment.

PBTS assume the largest burden of late effects from childhood cancer, with few effective solutions to address their lifelong challenges. Caregivers and families also experience stress and burden that can impact everyday functioning. Survivor's Journey Plus (SJ+) addresses this urgent need by offering a developmentally tailored, family-centered approach to improving social problem-solving, emotion-regulation, and metacognitive skills in PBTS, while offering strategies to reduce caregiver depression and family impact.

Our overarching objectives are to: 1) to refine the existing program based on feedback from patient advocates and establish usability and accessibility; 2) examine the efficacy of SJ+ in improving global QoL, internalizing symptoms, and EF skills in adolescent/emerging adult PBTS; and 3) examine the efficacy of SJ+ in reducing caregiver depression and family impact. Importantly, we will consider improvements in both patient-reported and performance-based outcomes. We will conduct a two-site, two-arm pilot RCT (n = 72) comparing SJ+ to an internet resource comparison (IRC) with outcomes assessed at baseline, treatment completion (~ 3 months post-baseline), and 6 months post-baseline.

SJ+ provides training in contextualized metacognitive strategies and communication skills to address common challenges (e.g., working memory, attention/planning, social communication) in the context of a broader social problem-solving framework. It is predicated on more than two decades of research with pediatric brain injury survivors, demonstrating its feasibility, acceptability, and efficacy among adolescents and young adults.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of a pediatric intracranial tumor
* tumor-directed treatment completed > 12 months ago (treatment included: surgery, radiation, or chemotherapy)
* lives with parent/guardian(s)
* language: English must be the primary spoken language in the home

Exclusion Criteria:

* history of tuberous sclerosis or neurofibromatosis
* treatment < 12 months ago and/or treatment did not include surgery, radiation, or chemotherapy
* history of psychiatric hospitalization
* resides outside of the family home
* history of autism, reactive attachment disorder, psychosis, or other psychiatric diagnoses/conditions associated with significant risk of harm to self or others per caregiver
* English is not the primary language spoken in the home

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Pediatric Quality of Life Inventory Total Scale Score change | From baseline to 6 months post-baseline
  Minimum score of 0, maximum score of 100. A higher score indicates better Health-Related Quality of Life, which is considered better.
Goal Attainment Scaling | From baseline to 6 months post-baseline.
  Method to establish individualized scales in order to quantify progress toward SMART personal goals.

SECONDARY OUTCOMES:
Behavior Rating Inventory of Executive Function, Second Edition T Scores change | From baseline to 6 months post-baseline
  Minimum T score of 0, maximum T score of 100. T scores at or above 70 are considered clinically elevated, which is considered worse.
Behavior Rating Inventory of Executive Function, Second Edition-Adult Version T Scores change | From baseline to 6 months post-baseline
  Minimum T score of 0, maximum T score of 100. T scores at or above 70 are considered clinically elevated, which is considered worse.
Patient-Reported Outcomes Measurement Information System change | From baseline to 6 months post-baseline
  Each measure has a range in score from 7 to 35 with higher scores indicating greater severity, which is considered worse.
Hospital Anxiety and Depression Scale change | From baseline to 6 months post-baseline
  Minimum score of 0, maximum score of 42. Higher scores mean greater levels of anxiety and depression, which is considered worse.
Strength & Difficulties Questionnaire change | From baseline to 6 months post-baseline
  Minimum score of 0, maximum score of 40. Higher scores mean greater levels of difficulties, which is considered worse.

CONTACTS AND LOCATIONS:
Overall Officials: Shari L Wade, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (2):
- United States (2):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No
The Dept of Defense will not need to see individual participant data from our study.